CLINICAL TRIAL: NCT00132132
Title: Type 2 Diabetes and Obesity Pediatric Prevention Project
Brief Title: Study of Impact of Behavioral Intervention- Exercise, Nutrition, Education- on Body Mass Index (BMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00203 (number assigned by IRB)
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: BMI; obesity; behavioral intervention; longterm randomized controlled trial; exercise; empowerment; nutrition
MeSH Terms: conditions — Obesity; Motor Activity; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This is a long term randomized controlled study looking at the effect of a Behavioral program on BMI in a population 10-20years old with a BMI greater than or equal to 85%. The intervention is a Behavioral education program which meets monthly for 4 hour session and includes exercise, education, empowerment and incentives. Both groups are referred to a dietician. The primary outcome is change in BMI and the secondary outcome is improvement in fasting metabolic parameters (lipid panel, insulin, glucose).
  Interventions: Behavioral: Behavioral education program
- Standard of Care/Control (No Intervention): Education on physical activity and nutrition in a primary care office setting

INTERVENTIONS:
Behavioral: Behavioral education program — Monthly 4 hr session which incorporates: exercise, empowerment, education, and incentives
  Arms: Intervention

SUMMARY:
This study will evaluate the impact a behavioral intervention can have on BMI. The researchers anticipate the intervention group will experience a decrease in BMI of approximately five points. The intervention group will be compared to a control group. This is a long term, randomized, controlled study. The behavioral intervention is conducted during a four hour monthly session. The behavioral intervention includes: exercise, education on medical aspects and nutrition, and empowerment.

DETAILED DESCRIPTION:
This is a long term randomized controlled trial, looking at the impact of a behavioral intervention on BMI,in participants ages 10-20 with a BMI > 85%.

The intervention group will:

* have baseline and follow up blood work (fasting insulin, glucose, lipid panel)
* have baseline and follow up BMI, blood pressure measurements
* see a dietician-minimum of three visits during study
* attend monthly, four hour sessions. These sessions include:

  1. registration-monitoring of choices of liquid intake using standardized models, monitoring of sedentary behaviors-hours watching television, computer, video games, monitoring of heart rate at baseline and after exercise, monitoring of METs (metabolic equivalents), motivational interviewing, monitoring of exercise abilities (endurance, agility, curl ups, balance, power)
  2. one hour of exercise (including strength training)
  3. educational lectures on nutrition and the medical aspects of obesity and Type 2 diabetes epidemic
  4. projects/games
  5. empowerment tools such as leading exercises and presenting food labels for discussion

The control group will have:

1. baseline and follow up blood work (fasting insulin, glucose, lipid panel)
2. baseline and follow up BMI and blood pressure measurements
3. visits to dietician (minimum of three visits during study)
4. standard education on nutrition and exercise given during office visit with primary care doctor

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-20 years
* BMI>85%

Exclusion Criteria:

* Endocrine disorder
* On psychotropic medications

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Gonzalez, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- Caritas St. Elizabeth's Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Program: This is a long term randomized controlled study looking at the effect of a Behavioral program on BMI in a population 10-20years old with a BMI greater than or equal to 85%. The intervention group attends a monthly 4 hour session which incorporates exercise, education, empowerment and incentives. Both groups are referred to a dietician. The primary outcome is change in BMI and the secondary outcome is improvement in fasting metabolic parameters (lipid panel, insulin, glucose).
- Standard of Care/Control: Standard of Care/control group received visits to the primary care provider and a referral to a nutritionist
Period: Overall Study
Arm/Group | Behavioral Program | Standard of Care/Control
Started | 15 | 15
Completed | 8 | 13
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Program | Standard of Care/Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI (Body Mass Index)
Time Frame: Baseline, 12-15 months
Population: Per protocol analysis: subjects who attended at least one intervention session in addition to their final assessment
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Groups:
- Intervention Group: The intervention group attended monthly, 4 hour sessions for one year
- Standard of Care/Control Group: The Standard of Care/Control group received visits to primary care provider and referral to nutritionist
Arm/Group | Intervention Group | Standard of Care/Control Group
Number analyzed (Participants) | 8 | 13
kg/m^2
  Unadjusted per-protocol change in BMI | -0.74 [-2.21 to 0.72] | 1.33 [0.18 to 2.48]
  Adjusted for age per-protocol change in BMI | -0.18 [-1.40 to 1.04] | 0.98 [0.04 to 1.93]
  Adjusted for age/paternal education change in BMI | -0.37 [-1.19 to 0.44] | 1.28 [0.59 to 1.97]
Statistical Analysis 1: Comparison: Intervention Group vs Standard of Care/Control Group; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; This analysis is the per protocol unadjusted value
Statistical Analysis 2: Comparison: Intervention Group vs Standard of Care/Control Group; Test type: Superiority or Other; p = 0.14, t-test, 2 sided; Age adjusted per protocol
Statistical Analysis 3: Comparison: Intervention Group vs Standard of Care/Control Group; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Per protocol adjusted for age and paternal education. Given the small number of participants with complete data, this model may be overfit

2. Primary Outcome: Percentage of Participants With BMI Reduction
Time Frame: Baseline, 12-15 months
Population: Per protocol
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Standard of Care/Control Group
Number analyzed (Participants) | 8 | 13
percentage of participants | 75 | 23
Statistical Analysis 1: Comparison: Intervention Group vs Standard of Care/Control Group; Test type: Superiority or Other; p = 0.02, Chi-squared

ADVERSE EVENTS:
Arm/Group | Behavioral Program | Standard of Care/Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
A limitation of the study is the lost to follow up. However, our rate of lost to follow up is comparable to rates seen in similar studies in this field

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes